CLINICAL TRIAL: NCT03691038
Title: Comparison of Conventional Flexible Dose Regimen of Pregabalin and New Flexible Dose Regimen of Pregabalin Using Low Dose: A Randomized Controlled Trial
Brief Title: Comparison of Conventional Dose Regimen and New Dose Regimen of Pregabalin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants couldn't be enrolled due to complain of frequent visit.
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoung-Ho Ryu, MD, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-08-013
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Pain, Neuropathic
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin 75mg bid (Active Comparator): The patients who were prescribed according to the conventional flexible dose regimen
  Interventions: Drug: Pregabalin 75mg bid
- pregabalin 25mg,50mg (Experimental): The patients who were prescribed according to the new flexible dose regimen.
  Interventions: Drug: Pregabalin 25mg, 50mg

INTERVENTIONS:
Drug: Pregabalin 75mg bid — Through the study period, Incremental protocol follows the conventional dose regimen starting pregabaline 75mg bid.
  Other Names: Conventional regimen
  Arms: Pregabalin 75mg bid
Drug: Pregabalin 25mg, 50mg — Through the study period, Incremental protocol follows the new dose regimen starting pregabalin 25mg, 50mg
  Other Names: New regimen
  Arms: pregabalin 25mg,50mg

SUMMARY:
The purpose of this study is to propose a new flexible dose regimen starting from 75mg using the low dose pregabalin 25 mg and 50 mg comparing the side effect and compliance with the conventional flexible dose regimen staring from 150mg using the pregabalin 75mg.

DETAILED DESCRIPTION:
Pregabalin has been shown to be effective as a first-line medication for neuropathic pain but it appears to have several side effects such as dizziness, drowsiness, and edema, which lowers compliance with medications. A way to reduce side effects is the flexible dose regimen, which reaches the target dose to treat the drug. The proposed flexible dose regimen is a regimen that begins with twice the prevalence of 75 mg. However, dizziness is the most common side effect up to 20% in conventional flexible dose regimen. Therefore, the aim of this study was to propose a new flexible regimen starting at a dose less than the existing dose and to compare compliance with pregabaline according to both methods

ELIGIBILITY:
Inclusion Criteria:

* Pain score NRS ≥3 Patients complaining of neuropathic pain (except neuropathic pain due to chemotherapy)
* Adult patients aged 19 to 85 years
* Patients who pre-agreed to the study

Exclusion Criteria:

* Patients complaining of severe pain (NRS ≥ 8)
* Creatinine clearance of <30 mL / min, the liver was more than 3 times normal
* Patients complaining of dizziness, patients with definite orthostatic hypotension
* Pregnant or lactating patients
* Patients who previously experienced side effects after administration pregabalin.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
discontinuation of medication | After 7 weeks of prescription
  the portion of patients discontinuing medication

CONTACTS AND LOCATIONS:
Overall Officials: Sung Hyun Lee, MD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No